CLINICAL TRIAL: NCT02381834
Title: Evaluation of a Novel Midstream Urine Collection Technique for Infants in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Eastern Ontario (Other)
Responsible Party: Principal Investigator, Tighe Crombie, Principal Investigator, Children's Hospital of Eastern Ontario
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14/190X
Record Dates: First submitted 2015-03-03; First posted 2015-03-06 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Urinary Tract Infection
Keywords: Urine Specimen Collection; Infant; Neonate; Bacterial Infection
MeSH Terms: conditions — Urinary Tract Infections; Bacterial Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bladder stimulation technique (Experimental): This is a two-person technique. A health care aide or nurse (RN) begins by holding the infant under the axillae with its legs dangling. A second RN or physician then performs bladder stimulation by gentle finger tapping on the lower abdomen in the midline just above the pubic symphysis at a frequency of 100 taps/min. If this is unsuccessful after 30 seconds, lower back stimulation in the lumbar paravertebral zone is performed by light massage in a circular motion using both thumbs. This too is performed for 30 seconds maximum. These two manoeuvres are repeated in succession, for a maximum of 5 minutes total, until urination occurs. Unsuccessful attempts at midstream urine collection will be followed by further feeding/fluid administration and bladder catheterization.
  Interventions: Procedure: Bladder stimulation technique

INTERVENTIONS:
Procedure: Bladder stimulation technique

SUMMARY:
Urinalysis and urine culture are commonly employed laboratory tests in the Emergency Department (ED), particularly for the purposes of investigating febrile infants in whom bacterial etiologies must be ruled out. The standard of care for obtaining sterile urine specimens in this age group remains transurethral bladder catheterization, an invasive procedure that is painful and has the potential for causing specimen contamination and iatrogenic urinary tract infection (UTI). A recent study by Herreros Fernández et al (2013) described a novel bladder stimulation technique for newborns that facilitates midstream urine collection. The success rate for this procedure was 86.3%. It remains unknown however as to whether this technique is reproducible amongst infants who present to the ED with a potentially greater severity of illness. The primary objective of this study is to determine the success rate of this technique in children ≤ 90 days old in the ED.

DETAILED DESCRIPTION:
Two persons (at least one trained nurse [RN] or physician [MD] and/or one health care aid [HCA]) will be required to perform the procedure, one of whom will also measure the time between critical steps of the protocol using a stopwatch. The technique involves a combination of fluid administration and non-invasive bladder stimulation manoeuvres that include gently finger tapping the abdomen with or without lower back massage.

The first step involves bottle or breastfeeding each infant with an amount of milk that is appropriate for its weight and age. Breastfed babies that have no history of poor feeding will be fed ad libitum. Those that feed poorly will be encouraged to supplement the feed with either expressed breast milk or formula at the discretion of the parent/guardian. Formula fed infants will receive a 10 ml feed on the first day of life, increasing by 10 ml per day of age to a maximum of 70 ml per feed. For infants greater than 7 days old, 25 ml/kg will be administered per feed. Babies that demonstrate mild clinical dehydration and/or fail attempts at oral feeding may, at the discretion of the most responsible physician (MRP), have a peripheral intravenous (IV) catheter placed and receive a fluid bolus of 0.9% normal saline up to a maximum of 10-20 ml/kg given over 20-25 minutes. Infants will not be excluded if they do not feed well.

Approximately 20 minutes after the feeding or IV fluid bolus, the infant's genitals will be cleaned in a sterile technique using 0.05% chlorhexidine. Non-pharmacological analgesia, as achieved with a soother and/or 24% sucrose will be offered to prevent or lessen crying.

The second major step of the technique involves holding the infant under the axillae with their legs dangling safely above the crib mattress. An RN or MD then begins bladder stimulation by gently finger tapping on the lower abdomen in the midline just above the pubic symphysis at a frequency of 100 taps per minute. If this step is unsuccessful after 30 seconds, the RN/MD will then stimulate the lower back in the lumbar paravertebral zone by lightly massaging the area in a circular motion using both thumbs. This too will be performed for a maximum of 30 seconds. The two stimulation manoeuvres will be repeated in succession (up to a maximum of 5 minutes, or 5 cycles) until micturition occurs and a midstream urine sample can be caught in a sterile container.

Infants who spontaneously urinate after cleaning, but prior to bladder stimulation, will have their clean catch urine sent to the lab. These cases will be considered successful "non-invasive" attempts.

Infants who fail to produce urine will have further feeding/fluid administration and bladder catheterization at the discretion of the MRP.

ELIGIBILITY:
Inclusion Criteria:

* Age ≤ 90 days
* Ped-CTAS (Canadian Pediatric Triage and Acuity Scale) Level = 2-5
* Urine specimen required for culture and/or urinalysis at the discretion of the most responsible physician (MRP) or as part of a nurse-initiated medical care directive

Exclusion Criteria:

* Age > 90 days
* Ped-CTAS Level = 1 (i.e. critically ill patient)
* Moderate to severe dehydration
* Significant feeding issues (e.g. suspected pyloric stenosis)
* Burn/infection/injury over site of bladder stimulation
* Previous enrollment

Max Age: 90 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2015-03; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients for whom the technique is successful for urine collection within 5 minutes (success being defined as the collection of an adequate sample volume [≥ 1 mL] for urinalysis and urine culture testing) | 5 minutes

SECONDARY OUTCOMES:
Proportion of contaminated samples (contamination being defined as growth of ≥ 2 microorganisms or growth of a single type of non-uropathogenic organism) | 24 hours
Length of bladder stimulation time (minutes) required for successful urine collection. | 5 minutes
Length of time (minutes) required to complete the full study protocol (from initiation of feeding/IV fluid administration to completed urine collection) | 1 hour
Patient distress as perceived by parent/guardian, measured using a 10 cm Visual Analog Scale (VAS). | 5 minutes
Components of satisfaction relating to the procedure for the parent/guardian and the Registered Nurse (RN) or Medical Doctor (MD) performing the procedure. | 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Tighe Crombie, MD, Principal Investigator — Children's Hospital of Eastern Ontario; Amy C Plint, MD, Principal Investigator — Children's Hospital of Eastern Ontario; Robert Slinger, MD, Principal Investigator — Children's Hospital of Eastern Ontario
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada